CLINICAL TRIAL: NCT01804881
Title: Effect of Beyond the Fork on Chronic Disease Self-management: a Pilot RCT
Brief Title: Effect of Managing Problematic Eating Behaviours With Dietary Management on Chronic Disease Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto Practice Based Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0225
Record Dates: First submitted 2013-03-02; First posted 2013-03-05 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-09

CONDITIONS: Hypertension; Type 2 Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Group program using Craving Change(tm) material was the intervention for dietary counseling, 6 group sessions
  Interventions: Behavioral: Lifestyle counseling
- Wait list control (Placebo Comparator): Wait list, offered group program using Craving Change(tm) material at end of study
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — Six week program to address problematic eating
  Other Names: Group program using Craving Change(tm) material

SUMMARY:
Dietary management is an integral aspect of self care for many chronic diseases. Craving Change™ is a standard program already offered at many Family Health Teams (FHT) to patients interested in being more mindful of their food choices. The program helps patients understand why they have difficulty with modifying behaviours associated with diet, addresses the impact of emotion on eating behaviour and provides affect regulation strategies. Existing literature shows that emotion has a strong effect on food choice and that emotion regulation can lead to improvements in food choice. Craving Change™, however, is currently not selectively offered at FHTs to patients deemed to be at higher risk of cardiovascular disease and has not been evaluated in that context. For this study, we propose to 1) Selectively target patients at higher cardiometabolic risk; and 2) Evaluate an effect of the program (as modified to address chronic diseases) through a pilot Randomized Controlled Trial (RCT). If found to be effective, the modified Craving Change™ program, called "Beyond the Fork: A health-centred approach to managing chronic disease", could be broadly implemented within Family Health Teams.

DETAILED DESCRIPTION:
This study is specifically focusing on Diabetes Mellitus Type 2 and Hypertension as these are chronic conditions in which dietary management is not only an integral part of managing the condition, but can also be a major factor in poor outcomes. Many of the current approaches and interventions used for treating these conditions provide patients with information about "what" eating behaviours to change and "how" to change them, such as through DEP (Diabetes Education Program) and CDSM (Chronic Disease Self-Management, aka Stanford).

The new intervention proposed in this study will be primarily based on material from the Craving Change™ program; the focus of which is to provide patients with an understanding of "why" it is difficult to change problematic eating behaviours. The new information that will be added is specific to chronic disease management. The original Craving Change™ program provides patients with information about how the environment, the physical body and emotional reactions can contribute to problematic eating behaviours thus increasing difficulty in changing those behaviours. The Craving Change™ program also provides patients with tools for overcoming the identified obstacles from the environment, physical body and emotional reactions in order to facilitate behaviour change. Patients who have a diagnosis of Diabetes Mellitus Type 2 and/or Hypertension and who are poorly controlled, are often required to make dietary changes to improve those conditions and often struggle to make the necessary dietary behaviour changes. By providing these patients with a behavioural intervention that uses the main components of the Craving Change™ program along with additional information specific to chronic disease management, the overall aim is to help patients improve control over the chronic condition with which they have been diagnosed.

As this is a feasibility study, the main goal is to determine if patients who are diagnosed with chronic disease(s) can be recruited successfully, stay in the program and experience a change in their perceptions of eating behaviours as a result of learning various strategies offered in the program. Specifically, this study is focusing on whether the strategies learned improve emotion regulation, which in turn could facilitate behaviour change. Our primary outcome measure is the EEQ ("Emotional Eater Questionnaire"); which is a validated 10 item questionnaire measuring the degree of interaction between emotion and food choice.

This study is a Randomized Control Trial. The setting is 3 Family Health Teams in the Greater Toronto Area. Eligibility criteria includes rostered status to the Family Health Team, no previous participation in a program using Craving Change™, diagnosis of Diabetes Mellitus Type 2 and/or Hypertension, and 2 of 3 high A1c / BP / LDL. Patients are identified using Electronic Medical Records (EMRs) and those patients meeting criteria are sent an EEQ via mail. Patients consenting to participation are invited to intake at which blood pressure (BP), height/weight/waist circumference (ht/wt/wc) is measured and patients are randomized to immediate participation in the program or to wait list control. After 6 weeks EEQ is re-administered, and BP, ht/wt/wc is measured again.

ELIGIBILITY:
Inclusion Criteria:

All participants must meet the following criteria to be included in the study:

* able to consent
* currently rostered to a physician in one of the three participating FHTs
* have never attended a program using Craving Change™ material
* live with Hypertension and/or Type 2 Diabetes
* and meet at least 2 out of 3 of the following criteria: A1C (last) >7.5% Systolic BP (last) > 140 LDL (last)> 4 (in non-diabetics) or >2 (for diabetics)

Exclusion Criteria:

* Physician opted out of the study, these patients will not be approached
* Participant does not consent
* Participant already attended Craving Change™ or a program using Craving Change™ material in the past
* Participant does not speak English

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danuta Southgate, MSW, RSW, Principal Investigator — North York Family Health Team
Locations (1):
- North York Family Health Team, Toronto, Ontario, Canada

REFERENCES:
- [Background] Evers C, Marijn Stok F, de Ridder DT. Feeding your feelings: emotion regulation strategies and emotional eating. Pers Soc Psychol Bull. 2010 Jun;36(6):792-804. doi: 10.1177/0146167210371383. Epub 2010 May 11. PMID 20460650
- [Background] Garaulet M, Canteras M, Morales E, Lopez-Guimera G, Sanchez-Carracedo D, Corbalan-Tutau MD. Validation of a questionnaire on emotional eating for use in cases of obesity: the Emotional Eater Questionnaire (EEQ). Nutr Hosp. 2012 Mar-Apr;27(2):645-51. doi: 10.1590/S0212-16112012000200043. PMID 22732995

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Counseling: Craving change group intervention for dietary counseling, 6 group sessions
  Lifestyle counseling: Six week program to address problematic eating
- Wait List Control: wait list, offered program based on craving change(tm) material at end of study
Period: Overall Study
Arm/Group | Lifestyle Counseling | Wait List Control
Started | 16 | 14
Completed | 11 | 10
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Counseling | Wait List Control | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (4.9) | 59.9 (7.5) | 61.7 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 14 | 30
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 31.2 (5.1) | 32.8 (5.1) | 32 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: The Change in EEQ (Emotional Eater Questionnaire) Score is the Primary Outcome Measure in This Study.
Description: The EEQ is a10-item validated questionnaire measuring the degree of interaction between food intake and emotion. Scores on a scale between baseline score and score after 6 weeks was measured.
  The EEQ is scored as follows:
  Values: Never = '0'; Sometimes = '1'; Generally = '2'; Always = '3' Score between 0-5: "You are a non-emotional eater. Score between 6-10: "You are a low emotional eater. Score between 11-20: "You are an emotional eater. Score between 21-30: "You are a very emotional eater. The participants completed the EEQ at baseline and it was scored. After 6 weeks the participants completed the EEQ again and it was scored again. The participants' baseline score was compared to the score at week 6. The goal was for scores to reduce. If participants' scores were higher at week 6, that could mean that the intervention was not successful. If the participants' scores were lower at week 6, that could mean that the intervention was successful.
Time Frame: 6 weeks
Population: Intention to Treat analysis
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Wait List Control: wait list, offered craving change program at end of study
Arm/Group | Lifestyle Counseling | Wait List Control
Number analyzed (Participants) | 13 | 12
Scores on a scale | -1.7 (2.6) | -3.2 (5.6)

2. Secondary Outcome: Change in Blood Pressure
Description: Blood Pressure was recorded at baseline and after 6 weeks. There are fewer participants recorded in this secondary outcome measure (11 and 10 vs.13 and 12 in previous, main, outcome measure) because some participants did not want to have blood pressure taken again.
Time Frame: 6 weeks
Population: Intention to Treat analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Lifestyle Counseling: Group intervention for dietary counseling, 6 group sessions
  Lifestyle counseling: Six week program to address problematic eating
- Wait List Control: wait list, offered group program at end of study
Arm/Group | Lifestyle Counseling | Wait List Control
Number analyzed (Participants) | 11 | 10
mm Hg
  Blood Pressure - Systolic | -3.3 (15.5) | -7.2 (15.3)
  Blood Pressure - Diastolic | 0.6 (6.6) | -6 (6.8)

3. Secondary Outcome: Change in Weight
Description: Weight was recorded at baseline and after 6 weeks. There are fewer participants recorded in this secondary outcome measure (11 and 10 vs.13 and 12 in previous, main, outcome measure) because some participants did not want to be re-weighed.
Time Frame: 6 weeks
Population: Intention to Treat analysis
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lifestyle Counseling | Wait List Control
Number analyzed (Participants) | 11 | 10
kg | -0.5 (0.9) | -0.87 (1.06)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lifestyle Counseling | Wait List Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
Small sample size is limitation and was affected by small number recruited due to some participants declining participation due to being unable to come in for the day/time group program was offered and some participants dropped out during the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No